CLINICAL TRIAL: NCT01985529
Title: A Controlled Study of Community-based Exercise Training in Patients With Moderate COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Shefalee Amin, Author, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 11-000175
Record Dates: First submitted 2013-11-01; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Enrollment in pulmonary rehabilitation
  Interventions: Other: Exercise
- Control (No Intervention)

INTERVENTIONS:
Other: Exercise
  Arms: Exercise

SUMMARY:
The effectiveness of clinic-based pulmonary rehabilitation in advanced Chronic Obstructive Pulmonary Disease (COPD) is well established, but few data exist for less severe patients treated in alternative settings. The purpose of this study was to investigate whether a novel, community-based exercise program was feasible and effective for patients with moderate COPD.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate COPD and self-reported exercise impairment

Exclusion Criteria:

* current smokers, pulmonary diseases other than COPD, use of supplemental oxygen, musculoskeletal disease that impaired exercise performance and unstable coronary artery disease or congestive heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Endurance | 12 weeks
  Change in endurance of physical activity was measured in seconds.

SECONDARY OUTCOMES:
Muscle Strength | 12 weeks
  Change in muscle strength was measures in pounds of weight lifted

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cooper, MD, Study Director — University of California, Los Angeles
Locations (1):
- UCLA, Westwood, Los Angeles, California, United States

REFERENCES:
- [Derived] Amin S, Abrazado M, Quinn M, Storer TW, Tseng CH, Cooper CB. A controlled study of community-based exercise training in patients with moderate COPD. BMC Pulm Med. 2014 Aug 4;14:125. doi: 10.1186/1471-2466-14-125. PMID 25088030